CLINICAL TRIAL: NCT00485563
Title: A Phase II Study of EC17 (Folate-hapten Conjugate) in Patients With Progressive Metastatic Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Changes in treatment paradigm resulted in a lower than expected rate of accrual.
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-FI-004
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Renal Cell Carcinoma
Keywords: Cancer; Vaccine; Phase 2; folate-hapten conjugate; Progressive; Metastatic; Experimental
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms; Neoplasm Metastasis | interventions — fluorescein isothiocyanate-keyhole limpet hemocyanin; GPI0100; Interleukin-2; aldesleukin; Interferon-alpha; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: EC90 (KLH-FITC) — 1.2mg in combination with adjuvant GPI-0100 administered subcutaneously (beneath the skin) weekly for 4 consecutive weeks during the first cycle of treatment, weekly for 2 consecutive weeks during the second cycle and once for each additional cycle.
  Other Names: Keyhole limpet hemocyanin fluorescein
Biological: GPI-0100 — 3.0 mg in combination with EC90 administered subcutaneously weekly for 4 consecutive weeks during the first cycle of treatment, weekly for 2 consecutive weeks during the second cycle and once for each additional cycle.
  Other Names: Saponin-based adjuvant
Drug: EC17 (Folate-FITC) — 0.3mg/kg administered subcutaneously 5 days per week (Monday through Friday) for 4 consecutive weeks for the first two treatment cycles and then 3 days per week (Monday, Wednesday, Friday) for 3 consecutive weeks for each additional cycle.
  Other Names: folate-fluorescein conjugate;; folate-hapten conjugate
Drug: Interleukin-2 — 7.0 MIU administered subcutaneously 3 times per week (Monday, Wednesday, Friday) for 4 consecutive weeks during the first 2 cycles of treatment, then 2.5 MIU administered subcutaneously 3 times per week (Monday, Wednesday, Friday) for 3 consecutive weeks for each additional cycle.
  Other Names: IL-2; Proleukin
Drug: Interferon-alpha — 3.0 MIU administered subcutaneously 3 times per week (Monday, Wednesday, Friday) for 4 consecutive weeks during the first 2 cycles of treatment, then 3.0 MIU administered subcutaneously 3 times per week (Monday, Wednesday, Friday) for 3 consecutive weeks for each additional cycle.
  Other Names: IFN-alpha; Intron-A

SUMMARY:
This is a Phase 2 clinical trial to collect data on tumor responses produced by folate-hapten conjugate therapy (vaccination with EC90 [KLH-FITC] and GPI-0100 adjuvant followed by treatment with EC17 (folate-FITC) in combination with low-dose cytokines in patients with progressive metastatic renal cell carcinoma. All patients will undergo imaging with the investigational imaging agent 99mTc-EC20 (FolateScan) during the screening period to confirm eligibility for the treatment portion of the clinical trial.

DETAILED DESCRIPTION:
Rationale: This is a Phase 2 study of folate-hapten conjugate therapy in combination with low-doses of the cytokines Interleukin-2 (IL-2) and Interferon-alpha (INF-alpha). Folate-hapten conjugate treatment consists of subcutaneous vaccinations with EC90, a compound designed to elicit an immune response (antibodies) to a dye called fluorescein (FITC), in combination with GPI-0100 adjuvant (a drug intended to improve antibody production). Vaccination is followed by treatment with EC17, a drug made by linking folate (a vitamin) with FITC. Experimental evidence has shown that the folate receptor is over-expressed in many human cancers, including renal cell carcinoma. It is expected that EC17 will attach to cancer cells through the folate receptor and that antibodies to FITC will recognize the cancer cell and mark it for destruction by the body's immune system. Two drugs, IL-2 and IFN-alpha, will be administered at low doses in combination with EC17 in order to boost the immune response. During the screening period, all potential patients will undergo imaging with 99mTc-EC20 (a technetium-based, folate- linked radiopharmaceutical [EC20]) for the purpose of identifying patients whose tumors express the folate receptor; the target of folate-hapten conjugate therapy. Prior to receiving EC90/GPI-0100 and EC17 therapy, patients must exhibit at least one tumor lesion that displays adequate uptake of 99mTc-EC20 during the imaging procedure.

ELIGIBILITY:
Inclusion Criteria:

* Must have a histologically confirmed diagnosis of renal cell carcinoma (clear cell or predominately clear cell component). Papillary histology may also be enrolled (maximum of 6 patients)
* Must be diagnosed with relapsed or Stage IV disease that is medically or surgically unresectable and that has progressed after systemic therapy, including at least one agent in the general class of kinase inhibitors (TKI not required for papillary histology)
* Must have measurable/evaluable metastatic disease sites that have not previously received radiotherapy and which does not require palliative intervention (at the time of enrollment). Patients with non-measurable/evaluable disease are ineligible
* Must have at least one tumor lesion that displays uptake of 99mTc-EC20
* Must be > than or = 18 years of age
* Women must either be 1)not of child-bearing potential of 2)have a negative serum pregnancy test within 7 days prior to commencing treatment with investigational agents
* Must have completed prior cytotoxic chemotherapy, radiotherapy, immunotherapy or experimental therapy 30 or more days prior to study enrollment, and recovered (or returned to baseline) from associated acute toxicities. This restriction excludes palliative radiotherapy.
* Must have an ECOG score less than or equal to 2
* Must have adequate hematologic, renal, and heptic function

Exclusion Criteria:

* Must not have a history of severe hypersensitivity (grade 3 - 4 allergic reaction) to fluorescein, radiological contrast agent, cytokines, or have received fluorescein within 30 days of the study
* Must not have medical conditions that preclude the use of IL-2 or IFN-α.
* Must not be pregnant or breast-feeding
* Must not be currently undergoing chemotherapy, anticancer hormonal therapy, and/or therapy with immunosuppressant agents
* Must not be currently receiving bisphosphonates such as Zometa® (unless started > four weeks prior to treatment with EC90/GPI-0100, in which case they can be continued)
* Must not have any concomitant malignancy with the exception of basal cell or squamous cell carcinoma of skin
* Must not have radiographically documented evidence of current brain metastases, a history of stem cell transplant, immunodeficiency, and/or a medical or psychiatric illness (that in the investigator's opinion, would prevent adequate compliance with study therapy or evaluation of the endpoints)
* Must not have been administered another radiopharmaceutical that would interfere with the assessment of 99mTc-EC20
* Must not be unable to tolerate conditions for radionuclide imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Response Rate - the proportion of subjects with objective response based on RECIST criteria | A minimum of 13 weeks (time to first follow-up CT)

SECONDARY OUTCOMES:
To assess the safety and tolerability of folate-hapten conjugate therapy | Duration of study drug administration + 30 days
Time-to-progression, response duration, overall survival time observed after folate-hapten conjugate therapy and ECOG performance status | Up to 2 years following completion of therapy
To assess the safety and tolerability of 99mTc-EC20 | Duration of study drug administration + 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Messmann, MD, MHS, BSc, Study Director — Endocyte
Locations (3):
- United States (3):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Methodist Hospital Research Institute, Houston, Texas